CLINICAL TRIAL: NCT03886051
Title: Assessment of Effect of Orthodontic Treatment on the Stability of Pre-Orthodontic Recession Coverage by Connective Tissue Graft. A Randomized Controlled Clinical Trial
Brief Title: Effect of Orthodontic Treatment on the Stability of Pre-Orthodontic Recession Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: perioloveleena
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Connective Tissue Graft before Orthodontic treatment
  Interventions: Procedure: Connective Tissue Graft before Orthodontic treatment
- control group (Active Comparator): Orthodontic treatment only
  Interventions: Procedure: Orthodontic treatment only

INTERVENTIONS:
Procedure: Connective Tissue Graft before Orthodontic treatment — Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage will be done using sub - epithelial connective tissue graft. Orthodontic treatment will be 3 months following the grafting procedure.
  Arms: test group
Procedure: Orthodontic treatment only — Scaling and root planing will be performed and after resolution of periodontal inflammation, orthodontic treatment will be initiated.
  Arms: control group

SUMMARY:
This study attempts to assess the effect of orthodontic treatment on the stability of pre-orthodontic recession coverage by connective tissue graft- a randomized controlled clinical trial and thus facilitate better evidence based treatment protocol.

DETAILED DESCRIPTION:
Gingival recession is the location of the gingival margin apical to the cemento-enamel junction. The consequences of gingival recession range from impairment of esthetics, development of dentin hypersensitivity, root caries and an especially high incidence of non-carious cervical lesions.

The etiology of gingival recession is held to be multifactorial with various predisposing and precipitating factors recognized. The most commonly implicated risk factors include bone dehiscence/fenestration, tooth malposition (especially facially positioned teeth), thin gingival phenotype, the narrow width of keratinized gingiva, frenum pull, the presence of gingival inflammation, overzealous toothbrushing, and faulty dental restorations. Apart from these, certain types of orthodontic tooth movements are also assumed to precipitate gingival recession although conclusive evidence in support of this postulation is still needed and if indeed true, the precise underlying mechanism still unclear.

Most of the studies have focused on the contribution of orthodontic treatment induced incisor proclination (outside the dentoalveolar envelope) as a causative factor for the development of gingival recession and the findings have been indecisive. While some studies support this premise, others have observed no such correlation. Correspondingly, the issue of periodontal intervention in order to prevent development and/or progression of gingival recession in patients scheduled for orthodontic treatment remains unclear. One approach supports performing gingival augmentation prior to initiation of orthodontic tooth movement. The basis for this approach rests in the concept of the importance of the minimum amount of attached gingiva needed for dissipating forces of muscle pull, unattached mucosa and masticatory stresses and facilitation of patient performed oral hygiene procedures. Esthetic improvement, management of dentinal hypersensitivity and prevention of root caries are other expected benefits specifically associated with performing root coverage surgery. Moreover, improvement of gingival tissue dimensions before orthodontic tooth movement is expected to prevent further deterioration of preexisting gingival recession and better withstand orthodontic forces. Therefore, this approach is typically a preventive one. However, supporters of the other perspective, i.e. waiting for gingival augmentation surgery until after orthodontic treatment is over believe that it is best to wait until the gingival recession develops into a pathological entity and becomes a real clinical problem warranting corrective treatment. In fact, they regard the aforementioned preventive approach as a sort of 'overtreatment' and therefore avoidable. There are also concerns expressed regarding the long-term stability of gingival marginal levels achieved with mucogingival surgery performed before orthodontic tooth movement. Based on the above discussion, it is apparent that there is wide subjectivity regarding clinical decision making in cases where orthodontic treatment is planned in patients displaying gingival recession. Currently, both the indications as well as the timing of carrying out root coverage procedures in patients scheduled for orthodontic treatment are not very well elaborated. A thorough search of the literature revealed a very modest level of evidence - one study with prospective and retrospective data collection and the other a retrospective study. In both the studies, gingival augmentation surgery was carried out before the orthodontic intervention. Therefore, a need is felt for conducting a well-designed research in order to dissipate the conflict of opinions existing over this vital clinical issue. The high prevalence of gingival recession among patients needing orthodontic treatment renders this question even more vital. The current study has thus been conceived and designed so as to help resolve this clinical decision making conundrum. In the proposed study, a comparative evaluation of clinical and radiographic parameters pre and post-orthodontic treatment in teeth with gingival recession between participants undergoing gingival recession coverage before the initiation of orthodontic tooth movement with participants not undergoing pre-orthodontic root coverage will be done. The root coverage procedure chosen is sub-epithelial connective tissue graft since it is recognized as the gold standard among all recession coverage surgical procedures.

The present prospective, analytical, randomized controlled clinical trial will be conducted in the Department of Periodontics and Oral Implantology in collaboration with Department of Orthodontics, Post Graduate Institute of Dental Sciences, Rohtak.

Systemically healthy individuals having slight crowding in the anterior region, with at least one tooth having a gingival recession in the same region.

Participants will be enlisted from the regular outpatient department of the Department of Periodontics and Oral Implantology, Department of Orthodontics and Department of Oral Medicine Diagnosis and Radiology after screening on the basis of inclusion and exclusion criteria as detailed above. All participants will be given an outline of the study design and all patient-specific considerations and concerns will be properly addressed. All participants will be required to provide written informed consent.

All patients enrolled in the study will be further randomly divided into the following two groups using computer-generated randomization table using block randomization of 4 and 6 by the random allocation software system.

1. Connective Tissue Graft before Orthodontic treatment (Test Group) - Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage will be done using subepithelial connective tissue graft. Orthodontic treatment will be initiated 3 months following the grafting procedure.
2. Orthodontic treatment only (Control Group) - Scaling and root planing will be performed and after resolution of periodontal inflammation, orthodontic treatment will be initiated.

Participants of both the groups will be regularly motivated and expected to maintain meticulous plaque control throughout the course of orthodontic treatment.

Full mouth scaling and root planning will be performed using ultrasonic instruments and hand instruments as needed. After administration of local anaesthesia, a partial-thickness flap will be reflected with a horizontal incision 2 mm away from the tip of the interdental papilla, and two vertical incisions will be made from the gingival margin of the line angles of adjoining teeth. These incisions would extend at least one tooth wider mesiodistally than the area of gingival recession. The incisions will be extended to the mucobuccal fold. A connective tissue graft will be obtained from the palate near the gingival margin of molars and premolars. The palatal wound will be sutured to obtain primary wound closure. The connective tissue graft will then be placed on the denuded root surface and sutured to the periosteum using resorbable sutures. The outer portion of the graft will be covered with the partial thickness flap, and sutures will be placed interdentally. This will be followed by placement of periodontal dressing. All the patients will be treated with the same fixed mechanotherapy. Oral hygiene motivation and maintenance will be done during the entire course of orthodontic treatment. Once the levelling and alignment (approximately 6-8 months) of teeth has been completed, parameters will be recorded for both test group and control group.

PRIMARY OUTCOME MEASURES A) Clinical:-

* Keratinized tissue width (KTW)
* Clinical attachment level(CAL)
* Recession depth (REC)
* Recession width
* Gingival Index(GI)
* Bleeding on Probing(BOP)

SECONDARY OUTCOME MEASURES A) Clinical:-

* Plaque Index
* Root Esthetic Score(RES)
* Probing pocket depth(PPD)
* Gingival Biotype/Phenotype
* Percentage of Root coverage
* Patient-based Evaluation of pain, hypersensitivity, and ease of oral hygiene maintenance by questionnaire and Visual Analogue scale for pain (VAS).

B) Radiographic:- Radiographic Investigations will be made at the start and at the end of the treatment using Customized bite blocks and parallel angle technique will be used to obtain Intra Oral periapical radiographs and measurements were calculated by using Image - J software.

DATA COLLECTION METHODS

Clinical:

Using University of North Carolina (UNC) 15 periodontal probe to measure PPD, CAL, BOP, gingival recession at 3 sites (mesiobuccal, distal buccal and midbuccal) per tooth and at 4 sites per tooth to measure PI and GI. The cemento-enamel junction will be used as a fixed reference point.

Radiographic:

Customized bite blocks and parallel angle technique will be used to obtain Intra Oral periapical radiographs and measurements were calculated by using Image- J software.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to the distribution of data. If found to be normal in distribution, intragroup comparison will be done by repeated ANOVA between different time points followed by paired T-test between two-time points and inter group comparison will be done by using Independent T-test between two groups. If it is in non-normal distribution, intragroup comparison will be done by Wilcoxon signed rank test and intergroup comparison will be done by Mann-Whitney U test. The Chi-square test will be applied to analyze categoric data. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-25 yrs.
* Anterior tooth displaying Miller's class III gingival recession.
* Gingival recession depth ≥ 2mm
* Arch length tooth material discrepancy ≤ 4 mm in anterior teeth which can be treated orthodontically without indication for planned extraction.
* At the time of enrollment, the patient not having trauma from occlusion.
* Presence of clinically identifiable cementoenamel junction.
* Patient demonstrating compliance for maintaining good oral hygiene after Phase I treatment.

Exclusion Criteria:

* Patient having any systemic illness (such as diabetes, hyperthyroidism, autoimmune diseases, etc.) that is known to affect the periodontium or outcome of periodontal treatment.
* Aggressive Periodontitis
* Patients taking medications such as corticosteroids or calcium channel blockers, which are known to interfere with periodontal wound healing or patients on long-term NSAIDS treatment.
* Patients allergic to medication (local anaesthetic, antibiotic, NSAID).
* Pregnant or lactating women.
* History of recent periodontal treatment within 6 months prior to the study.
* Teeth Displaying Miller's class III/class IV gingival recession.
* The presence of severe cervical abrasion, erosion or root caries that would require restoration and cervically restored teeth.
* Patients indicated for planned extraction during orthodontic treatment.
* Gingival recession in due to extrusion of the tooth.
* Mobile teeth.
* Non-vital tooth.
* Smokers and tobacco chewers.
* Patients with Oral Piercing.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
recession depth | approximate 14 months
  • Recession depth (REC) recorded in mm from the cementoenamel junction to the crest of the gingival margin at the deepest point

CONTACTS AND LOCATIONS:
Overall Officials: SHIKHA TEWARI, Study Director — Post Graduate institute of dental sciences ROHTAK,HARYANA,INDIA
Locations (1):
- Shikha Tewari, Rohtak, Haryana, India